CLINICAL TRIAL: NCT02250638
Title: A Prospective Longitudinal Study of CA 19-9 as an Aid in Monitoring Disease in Patients With Pancreatic Cancer
Brief Title: Longitudinal Pancreatic Cancer Study
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FDI-68
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2020-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and Plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: CA 19-9 Assay — Physicians use the CA 19-9 test results to manage their patients

SUMMARY:
To obtain sufficient specimens and correlating clinical data from a well-controlled prospective clinical trial collecting longitudinal specimens from subjects diagnosed with any stage of pancreatic cancer.

DETAILED DESCRIPTION:
The study objectives are described below:

1. Obtain serum and plasma specimens longitudinally collected from approximately 140 subjects diagnosed with pancreatic cancer and are about to or are currently undergoing treatment and follow-up. Specimens will be used to evaluate CA 19-9 assays, currently under development, as an aid for monitoring recurrence or progressive disease.
2. To store any remaining specimens for use in future cancer research and to evaluate as yet undetermined biomarkers for the development of IVDs, including additional CA 19-9 assays, for monitoring the course of disease and therapy in subjects diagnosed with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age≥ 18 years
* Histologic/pathologic confirmation of exocrine pancreatic cancer
* Any stage of disease: Newly diagnosed, stable, disease progression
* Any treatment time point: Treatment naïve, currently receiving or completed therapy for pancreatic cancer including active monitoring.
* Individuals with a history of malignant disease other than pancreatic cancer that was resected greater than 5 years ago and are currently in remission are eligible.
* Life expectancy greater than 6 months
* Able to understand and willing to provide informed consent

Exclusion Criteria:

* Males and females, age <18 years
* No histologic/pathologic confirmation of exocrine pancreatic cancer
* Life expectancy less than 6 months
* Any concurrent malignancy other than basal or squamous cell skin cancers or in-situ cervical cancer.
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 140 subjects will be enrolled in this study. Women and men greater than or equal to 18 years of age with a histologically/pathologically confirmed diagnosis of pancreatic cancer and a minimum of three serial blood draws collected at disease evaluation time points, as determined by the treating physician's standard of care, will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2014-05; Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
A Prospective Longitudinal Study of CA 19-9 as an Aid in Monitoring Disease in Patients with Pancreatic Cancer | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Diana Dickson, Study Director — Fujirebio Diagnostics, Inc.
Locations (7):
- United States (6):
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Harry & Jeanette Weinberg Cancer Institute, Baltimore, Maryland
  - Kansas City VA Center, Kansas City, Missouri
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - The Ohio State University, Columbus, Ohio
- GI Research Institute, Vancouver, British Columbia, Canada